CLINICAL TRIAL: NCT01090011
Title: A Phase Ib Open-label Clinical Trial of Continuous Once Daily Oral Treatment Using BIBW 2992 Plus Cetuximab (Erbitux®) in Patients With Non-small Cell Lung Cancer With Progression Following Prior Erlotinib (Tarceva®) or Gefitinib (Iressa®)
Brief Title: Trial of BIBW 2992 (Afatinib) + Cetuximab in Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1200.71; 2009-015911-42 (EudraCT Number: EudraCT)
Record Dates: First submitted 2010-03-10; First posted 2010-03-19 (Estimated); Results first posted 2014-07-21 (Estimated); Last update posted 2015-10-02 (Estimated); Status verified 2015-08

CONDITIONS: Carcinoma, Non-Small-Cell Lung
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Cetuximab; Afatinib

ARMS (2):
- combination arm (Experimental): patients to receive medium BIBW 2992 once daily plus biweekly cetuximab infusion at low, median and high dose level
  Interventions: Drug: Cetuximab; Drug: BIBW 2992
- sequential arm (Experimental): patients to receive BIBW 2992 once daily, upon progression add biweekly cetuximab
  Interventions: Drug: Cetuximab; Drug: BIBW 2992

INTERVENTIONS:
Drug: Cetuximab — BIBW 2992 medium dose plus high dose level of cetuximab
  Arms: combination arm
Drug: Cetuximab — BIBW 2992 medium dose monotherapy, upon progression, cetuximab high dose is added
  Arms: sequential arm
Drug: BIBW 2992 — BIBW 2992 medium dose plus high dose level of cetuximab
  Arms: combination arm
Drug: BIBW 2992 — BIBW 2992 medium dose monotherapy, upon progression, cetuximab high dose is added
  Arms: sequential arm

SUMMARY:
The primary objective of this trial is to determine the maximum tolerated dose (MTD) and recommended Phase II doses for the combination of BIBW 2992 and cetuximab in patients with non-small cell lung cancer and acquired resistance to erlotinib or gefitinib.

Overall safety, pharmacokinetics and anti-tumor activity for the combination of BIBW 2992 and cetuximab in patients with non-small cell lung cancer and acquired resistance to erlotinib, gefitinib or BIBW 2992 will be evaluated as secondary objectives.

Initially a standard, 3+3 dose escalation will be performed to determine the MTD of BIBW 2992 when administered together with cetuximab in patients with advanced non small cell lung cancer and acquired resistance to erlotinib or gefitinib.

Subsequently, the preliminary efficacy and safety of the identified MTD of cetuximab administered with BIBW 2992 will be explored in a combo arm via a further expansion of MTD cohort up to a total of 140 EGFR mutation positive NSCLC with acquired resistance to erlotinib/gefitinib.

Furthermore, the safety and preliminary anti-tumor activity of the combination therapy in EGFR mutant NSCLC patients who developed acquired resistance (AR) to BIBW 2992, will be assessed in a sequential arm. The sequential arm will use a two-stage design with an early stopping rule after 12 patients with acquired resistance to BIBW 2992 have received up to 5 courses of BIBW 2992 plus cetuximab. If no responses are seen in 12 patients during 5 courses of combination therapy, accrual in the sequential arm will stop. If 1 or more responses are observed, the sequential arm will expand up to about 40 patients.

ELIGIBILITY:
Inclusion criteria:

1. Pathologically or cytologically confirmed Stage IIIB/IV non-small cell lung cancer or recurrent disease following locoregional treatment
2. Either or both of the following:

1) A tumor which harbors an Epidermal Growth Factor Receptor (EGFR) -mutation known to be associated with drug sensitivity (i.e., G719X, exon 19 deletion, L858R, L861Q) from previous tumor biopsy or surgery. A tumor which harbors exon 20 insertion or de novo T790M mutation is eligible for the treatment in the sequential arm 2) Objective clinical benefit from treatment with an Epidermal Growth Factor Receptor Tyrosine Kinase Inhibitor (EGFR TKI) as defined by either

1. Documented partial or complete response (Response Evaluation Criteria in Solid Tumors, RECIST), or
2. Stable disease >=6 months as defined by RECIST in absence of radiographic progression after initiation of gefitinib or erlotinib; or stable disease/PR/CR >=12 weeks as defined by RECIST after initiation of BIBW 2992 3. Systemic progression of disease (RECIST v1.1) while on continuous treatment with erlotinib or gefitinib or BIBW 2992 within the last 30 days. Patients whose disease progresses only in the central nervous system (CNS) are not eligible 4. No intervening systemic therapy between cessation of gefitinib or erlotinib or BIBW 2992 and initiation of the treatment in the study 5. Adequate tumor-derived material such as fresh or archived tumor tissue or pleural fluid from malignant pleural effusion after disease progression on erlotinib/gefitinib/BIBW 2992 prior to the study entry must be made available for EGFR mutation analyses 6. Patients aged 18 years or older 7. Life expectancy of at least three (3) months 8. Eastern Cooperative Oncology Group (ECOG) performance score 0-2 9. Written informed consent that is consistent with ICH-GCP guidelines

Exclusion criteria:

1. Prior treatment with EGFR targeting antibodies; prior severe infusion reaction to a monoclonal antibody
2. Adverse events due to major surgery (at least 28 days after) or minor surgery not recovered to CTC grade 1 or less. Surgical wounds must be healing without clinical evidence of infection prior to study treatment to be eligible.
3. Radiotherapy less than two weeks prior to the start of the study treatment
4. Systemic chemotherapy, hormonal therapy, immunotherapy, or experimental or approved proteins/antibodies (except erlotinib/gefitinib/BIBW 2992) <=30 days before study treatment
5. Less than three days from prior treatment with gefitinib or erlotinib. Patients with adverse events related to gefitinib or erlotinib must recover to CTC AE grade 1 or less to be eligible. No need to stop BIBW 2992 before start of the study treatment for patient who progressed on BIBW 2992 from a separate clinical trial/treatment setting
6. Brain metastases, which are symptomatic. Patients with treated, asymptomatic brain metastases are eligible if there has been no change in brain disease status for at least four (4) weeks, no history of cerebral oedema or bleeding in the past four (4) weeks. Anticonvulsant therapy will be allowed if patient is stable on anticonvulsant treatment.
7. Other malignancies diagnosed within the past five (5) years (other than non melanomatous skin cancer, ductal carcinoma in situ and in situ cervical cancer)
8. Known pre-existing interstitial lung disease
9. Significant or recent acute gastrointestinal disorders with diarrhea as a major symptom e.g., Crohns disease, malabsorption, or Common Toxicity Criteria for Adverse Events (CTCAE) grade >2 diarrhea of any etiology
10. Women of childbearing potential (WOCBP), or men who are able to father a child, unwilling to use a medically acceptable method of contraception during the trial; pregnancy or breast-feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 171 (Actual)
Dates: Start 2010-03; Primary Completion 2013-01 (Actual); Study Completion 2014-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (6):
- United States (4):
  - 1200.71.1004 Boehringer Ingelheim Investigational Site, Aurora, Colorado
  - 1200.71.1003 Boehringer Ingelheim Investigational Site, New Haven, Connecticut
  - 1200.71.1001 Boehringer Ingelheim Investigational Site, New York, New York
  - 1200.71.1002 Boehringer Ingelheim Investigational Site, Nashville, Tennessee
- Netherlands (2):
  - 1200.71.2002 Boehringer Ingelheim Investigational Site, Amsterdam
  - 1200.71.2001 Boehringer Ingelheim Investigational Site, Groningen

REFERENCES:
- [Derived] Horn L, Gettinger S, Camidge DR, Smit EF, Janjigian YY, Miller VA, Pao W, Freiwald M, Fan J, Wang B, Chand VK, Groen HJM. Continued use of afatinib with the addition of cetuximab after progression on afatinib in patients with EGFR mutation-positive non-small-cell lung cancer and acquired resistance to gefitinib or erlotinib. Lung Cancer. 2017 Nov;113:51-58. doi: 10.1016/j.lungcan.2017.08.014. Epub 2017 Aug 31. PMID 29110849
- [Derived] Janjigian YY, Smit EF, Groen HJ, Horn L, Gettinger S, Camidge DR, Riely GJ, Wang B, Fu Y, Chand VK, Miller VA, Pao W. Dual inhibition of EGFR with afatinib and cetuximab in kinase inhibitor-resistant EGFR-mutant lung cancer with and without T790M mutations. Cancer Discov. 2014 Sep;4(9):1036-45. doi: 10.1158/2159-8290.CD-14-0326. Epub 2014 Jul 29. PMID 25074459

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 171 patients were entered and treated in the study.
Groups:
- Total Patients: All patients entered and treated. The objective of this study was to determine the maximum tolerated dose of Afatinib using a "3+3 Up-and-Down" trial design. Cohorts of three to six participants were entered (not randomized) sequentially into escalating dosage tiers of afatinib/cetuximab. The dose of cetuximab in successive cohorts was increased unless two or more of the six participants (of the current cohort) had dose limiting toxicity events.
Period: Overall Study
Arm/Group | Total Patients
Started | 171
Completed | 0
Not Completed | 171
Not completed — Progressive disease | 128
Not completed — Adverse Event | 32
Not completed — Protocol Violation | 1
Not completed — Refusal to start/continue medication | 5
Not completed — Other reason not defined above | 5

BASELINE CHARACTERISTICS:
Population: Treated set which includeed all patients enrolled in the trial who were documented to have taken at least one dose of study medication.
Arm/Group | Total Patients
Number analyzed (Participants) | 171
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.1 (10.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 119
  Male | 52

OUTCOME MEASURES:

1. Primary Outcome: The Primary Endpoint is the Occurrence of Dose Limiting Toxicity (DLT).
Description: A DLT was defined as an AE or laboratory abnormality that a) related to the study regimen; b) or met any of the following criteria:
  * CTCAE Grade 2 or higher decrease in cardiac left ventricular function
  * CTCAE Grade 2 diarrhea lasting for 7 or more days, despite appropriate use of standard anti-diarrheal therapy
  * CTCAE Grade ≥3 diarrhea despite appropriate use of standard anti-diarrheal therapy for at least 2 days
  * CTCAE Grade ≥3 nausea and/or vomiting despite appropriate use of standard anti-emetics for at least 3 days
  * CTCAE Grade ≥3 rash despite standard medical management
  * CTCAE Grade ≥3 fatigue lasting for more than 7 days
  * CTCAE Grade 4 hypomagnesaemia or Grade 3 hypomagnesaemia with clinical significant sequelae
  * All other toxicities of CTCAE Grade ≥3 (except alopecia, and allergic reaction) leading to an interruption of afatinib and/or cetuximab for more than 14 days until recovery to baseline or Grade 1, whichever was higher.
Time Frame: from day 1 treatment until progression or undue toxicity, up to 28 days
Population: Treated set for Cohort One. Cohort one was based on the data from the first treatment cycle where four patients received 'Afatinib 40+Cetuximab 250' and six patients received 'Afatinib 40+Cetuximab 500'.
Measure: Number; unit: participants
Groups:
- Combination Arm - Afa40+Ctx250: Combination Arm (includes the initial dose escalation and expansion cohort of upfront afatinib plus cetuximab in patients with Acquired Resistance (AR) to erlotinib or gefitinib)
  Afatinib 40 mg + cetuximab 250 mg/m2 (Afa40+Ctx250)
- Combination Arm - Afa40+Ctx500: Combination Arm (includes the initial dose escalation and expansion cohort of upfront afatinib plus cetuximab in patients with AR to erlotinib or gefitinib)
  Afatinib 40 mg + cetuximab 500 mg/m2 (Afa40+Ctx500)
Arm/Group | Combination Arm - Afa40+Ctx250 | Combination Arm - Afa40+Ctx500
Number analyzed (Participants) | 4 | 6
participants | 0 | 0

2. Secondary Outcome: Highest CTCAE Grade
Description: Safety of afatinib when administered together with cetuximab as indicated by intensity and incidence of adverse events, graded according to the U.S. National Cancer Institute (NCI) Common Toxicity Criteria for Adverse Events (CTCAE) Version (v) 3.0
Time Frame: From first drug administration to 28 days after discontinuation of drug intake up to 915 days
Population: Treated set. 32 patients in the Afa40-mono group had disease progression and were transitioned to treatment with Afa40+Ctx500. Thus the total of 203 patients (4+126+37+36) minus the 32 patients counted in both 'Afa-mono' and 'Afa40+Ctx500' treatments arms equals 171, the total number of patients started in participant flow section.
Measure: Number; unit: percentage of patients
Groups:
- Combination Arm - Afa40+Ctx250: Combination Arm (includes the initial dose escalation and expansion cohort of upfront afatinib plus cetuximab in patients with AR to erlotinib or gefitinib)
  Afatinib 40 mg + cetuximab 250 mg/m2 (Afa40+Ctx250)
- Sequential Arm - Afatanib Monotherapy (Afa40 Mono): Sequential Arm (includes patients who received afatinib monotherapy and upon progression the combination of afatinib and cetuximab at the Maximum Tolerated Dose (MTD) determined in the combination arm. Patients still needed to have met the criteria for AR to erlotinib or gefitinib)
  Afatinib 40 mg (Afa40 Mono)
- Sequential Arm - Combination Therapy (Afa40+Ctx500): Sequential Arm (includes patients who received afatinib monotherapy and upon progression the combination of afatinib and cetuximab at the MTD determined in the combination arm. Patients still needed to have met the criteria for AR to erlotinib or gefitinib)
  Afatinib 40 mg + cetuximab 500 mg/m2 (Afa40+Ctx500)
Arm/Group | Combination Arm - Afa40+Ctx250 | Combination Arm - Afa40+Ctx500 | Sequential Arm - Afatanib Monotherapy (Afa40 Mono) | Sequential Arm - Combination Therapy (Afa40+Ctx500)
Number analyzed (Participants) | 4 | 126 | 37 | 36
percentage of patients
  Patients with highest CTCAE Grade 1 | 0 | 0.8 | 10.8 | 2.8
  Patients with highest CTCAE Grade 2 | 25.0 | 26.2 | 24.3 | 19.4
  Patients with highest CTCAE Grade 3 | 50.0 | 54.0 | 48.6 | 52.8
  Patients with highest CTCAE Grade 4 | 25.0 | 4.0 | 5.4 | 8.3
  Patients with highest CTCAE Grade 5 | 0 | 15.1 | 10.8 | 16.7

3. Secondary Outcome: Frequency of Patients [N(%)] With Possible Clinically Significant Abnormalities for Selected Laboratory Parameters
Time Frame: From first drug administration to 28 days after discontinuation of drug intake up to 915 days
Population: as for outcome 2
Measure: Number; unit: percentage of patients
Groups:
- Sequential Arm - Afatanib Monotherapy (Afa40 Mono): Sequential Arm (includes patients who received afatinib monotherapy and upon progression the combination of afatinib and cetuximab at the MTD determined in the combination arm. Patients still needed to have met the criteria for AR to erlotinib or gefitinib)
  Afatinib 40 mg (Afa40 Mono)
Arm/Group | Combination Arm - Afa40+Ctx250 | Combination Arm - Afa40+Ctx500 | Sequential Arm - Afatanib Monotherapy (Afa40 Mono) | Sequential Arm - Combination Therapy (Afa40+Ctx500)
Number analyzed (Participants) | 4 | 126 | 37 | 36
percentage of patients
  Haemoglobin - low (N=4,124,35,35) | 0 | 12.9 | 20.0 | 2.9
  White blood cell ct. - low (N=4,124,35,35) | 0 | 3.2 | 0 | 2.9
  Neutrophils - low (N=4,124,35,35) | 0 | 4.0 | 0 | 2.9
  Sodium - low (N=4,124,35,35) | 0 | 5.6 | 0 | 2.9
  Potassium - low (N=4,124,35,35) | 0 | 5.6 | 2.9 | 5.7
  Potassium - high (N=4,124,35,35) | 0 | 4.0 | 0 | 0
  Calcium - low (N=4,124,35,35) | 0 | 6.5 | 8.6 | 5.7
  Calcium - high (N=4,124,35,35) | 0 | 1.6 | 0 | 0
  Magnesium - low (N=4,124,34,35) | 0 | 9.7 | 0 | 11.4
  AST/GOT, SGOT - high (N=4,123,35,35) | 0 | 3.3 | 0 | 2.9
  ALT/GPT, SGPT - high (N=4,123,35,35) | 0 | 11.4 | 0 | 8.6
  Alkaline phosphatase - high (N=4,124,35,35) | 25.0 | 4.8 | 2.9 | 5.7
  Blood urea nitrogen - high (N=missing,105,28,28) | 0 | 5.7 | 3.6 | 0
  Creatinine - high (N=4,123,33,35) | 0 | 2.4 | 0 | 0
  Creatinine clearance - low (N=4,123,33,35) | 0 | 3.3 | 0 | 2.9
  Bilirubin,total - high (N=4,124,35,35) | 0 | 4.8 | 2.9 | 5.7
  Sodium - high (N=4,124,35,35) | 0 | 0.8 | 0 | 0

4. Secondary Outcome: Frequency (%) of Patients With Adverse Events Leading to Dose Reduction
Time Frame: From first drug administration to 28 days after discontinuation of drug intake up to 915 days
Population: as for outcome 2
Measure: Number; unit: percentage of patients
Arm/Group | Combination Arm - Afa40+Ctx250 | Combination Arm - Afa40+Ctx500 | Sequential Arm - Afatanib Monotherapy (Afa40 Mono) | Sequential Arm - Combination Therapy (Afa40+Ctx500)
Number analyzed (Participants) | 4 | 126 | 37 | 36
percentage of patients | 25.0 | 37.3 | 13.5 | 22.2

5. Secondary Outcome: Frequency (%) of Patients With Adverse Events Leading to Treatment Discontinuation
Description: Frequency (%) of patients with adverse events leading to treatment discontinuation
Time Frame: From first drug administration to 28 days after discontinuation of drug intake up to 915 days
Population: as for outcome 2
Measure: Number; unit: percentage of patients
Arm/Group | Combination Arm - Afa40+Ctx250 | Combination Arm - Afa40+Ctx500 | Sequential Arm - Afatanib Monotherapy (Afa40 Mono) | Sequential Arm - Combination Therapy (Afa40+Ctx500)
Number analyzed (Participants) | 4 | 126 | 37 | 36
percentage of patients | 50.0 | 23.8 | 2.7 | 19.4

6. Secondary Outcome: Frequency (%) of Patients With Adverse Events Leading to Death
Time Frame: From first drug administration to 28 days after discontinuation of drug intake up to 915 days
Population: as for outcome 2
Measure: Number; unit: percentage of patients
Arm/Group | Combination Arm - Afa40+Ctx250 | Combination Arm - Afa40+Ctx500 | Sequential Arm - Afatanib Monotherapy (Afa40 Mono) | Sequential Arm - Combination Therapy (Afa40+Ctx500)
Number analyzed (Participants) | 4 | 126 | 37 | 36
percentage of patients | 0.0 | 15.1 | 10.8 | 16.7

7. Secondary Outcome: Frequency (%) of Patients With Related Serious Adverse Events
Description: Frequency (%) of patients with drug-related serious adverse events
Time Frame: From first drug administration to 28 days after discontinuation of drug intake up to 915 days
Population: as for outcome 2
Measure: Number; unit: percentage of patients
Arm/Group | Combination Arm - Afa40+Ctx250 | Combination Arm - Afa40+Ctx500 | Sequential Arm - Afatanib Monotherapy (Afa40 Mono) | Sequential Arm - Combination Therapy (Afa40+Ctx500)
Number analyzed (Participants) | 4 | 126 | 37 | 36
percentage of patients | 0.0 | 10.3 | 5.4 | 2.8

8. Secondary Outcome: Area Under the Concentration-time Curve (AUC) on Day 15 of Plasma Afatinib for the Combination Arm
Description: Area Under the Concentration-time Curve (AUC) of Afatinib in plasma at steady state over a uniform dosing interval tau (15 days) (AUCtau,ss) after oral administration of Afatinib and cetuximab combination therapy
Time Frame: Course 1, Visit 3 and 4, Day 15 and 16, Hours: -0:05,0,1,2,3,4,5,6,8, and 23:55
Population: Pharmacokinetic dataset (PKS)
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Combination Arm - Afa40+Ctx250 | Combination Arm - Afa40+Ctx500
Number analyzed (Participants) | 3 | 20
ng*h/mL | 1300 (21.8) | 935 (59.8)

9. Secondary Outcome: Concentration of Afatinib in Plasma for the Combination Arm
Description: Minimum measured concentration of Afatinib in plasma at steady state over 15 day dosing interval (Cmin,ss). Maximum measured concentration of Afatinib in plasma at steady state over 15 day dosing interval (Cmax,ss).
Time Frame: Course 1, Visit 3 and 4, Day 15 and 16, Hours: -0:05,0,1,2,3,4,5,6,8, and 23:55
Population: Pharmacokinetic dataset (PKS)
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Combination Arm - Afa40+Ctx250 | Combination Arm - Afa40+Ctx500
Number analyzed (Participants) | 3 | 24
ng/mL
  Cmin,ss,15 | 33.9 (19.6) | 24.4 (53.7)
  Cmax,ss,15 | 83.8 (19.8) | 52.3 (73.2)

10. Secondary Outcome: Peak-trough Fluctuation (PTF)
Description: Peak-trough fluctuation (PTF) of plasma afatinib for the combination arm. PTF = 100*(Cmax-Cmin)/Caverage where Caverage = AUC/time, where time equals 24 hours.
Time Frame: Course 1, Visit 3 and 4, Day 15 and 16, Hours: -0:05,0,1,2,3,4,5,6,8, and 23:55
Population: Pharmacokinetic dataset (PKS)
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: % of average concentration
Arm/Group | Combination Arm - Afa40+Ctx250 | Combination Arm - Afa40+Ctx500
Number analyzed (Participants) | 3 | 20
% of average concentration | 91.6 (15.9) | 73.8 (55.2)

11. Secondary Outcome: t1/2,ss
Description: Terminal half-life of Afatinib in plasma at steady state (t1/2,ss)
Time Frame: Course 1, Visit 3 and 4, Day 15 and 16, Hours: -0:05,0,1,2,3,4,5,6,8, and 23:55
Population: Pharmacokinetic dataset (PKS)
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h
Arm/Group | Combination Arm - Afa40+Ctx250 | Combination Arm - Afa40+Ctx500
Number analyzed (Participants) | 3 | 21
h | 22.4 (24.5) | NA (NA) — No descriptive statistics calculated due to insufficient number of participants with data

12. Secondary Outcome: MRTpo,ss
Description: mean residence time of Afatinib in the body at steady state after oral administration (MRTpo,ss) for 15 days
Time Frame: Course 1, Visit 3 and 4, Day 15 and 16, Hours: -0:05,0,1,2,3,4,5,6,8, and 23:55
Population: Pharmacokinetic dataset (PKS)
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h
Arm/Group | Combination Arm - Afa40+Ctx250 | Combination Arm - Afa40+Ctx500
Number analyzed (Participants) | 3 | 20
h | 32.6 (23.4) | NA (NA) — no descriptive statistics calculated due to insufficient number of participants with data

13. Secondary Outcome: CL/F,ss,15
Description: Apparent clearance of afatinib in plasma at steady state after extravascular multiple dose administration (CL/F,ss)
Time Frame: Course 1, Visit 3 and 4, Day 15 and 16, Hours: -0:05,0,1,2,3,4,5,6,8, and 23:55
Population: Pharmacokinetic dataset (PKS)
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mL/min
Arm/Group | Combination Arm - Afa40+Ctx250 | Combination Arm - Afa40+Ctx500
Number analyzed (Participants) | 3 | 20
mL/min | 511 (21.8) | 713 (59.8)

14. Secondary Outcome: Vz/F,ss
Description: Apparent volume of distribution during the terminal phase λz at steady state following extravascular administration (Vz/F,ss) for 15 days
Time Frame: Course 1, Visit 3 and 4, Day 15 and 16, Hours: -0:05,0,1,2,3,4,5,6,8, and 23:55
Population: Pharmacokinetic dataset (PKS)
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L
Arm/Group | Combination Arm - Afa40+Ctx250 | Combination Arm - Afa40+Ctx500
Number analyzed (Participants) | 3 | 21
L | 991 (44.8) | NA (NA) — no descriptive statistics calculated due to insufficient number of participants with data

15. Secondary Outcome: Predose Plasma Concentrations of Afatinib for the Combination Arm
Description: Predose plasma concentrations (Cpre,ss) of Afatinib at Course 1, Visit 2, 3, 4 and 5, at Course 2, Visit 1 and 2 and at Course 3, Visit 1.
Time Frame: Up to 57 days
Population: Pharmacokinetic dataset (PKS)
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Combination Arm - Afa40+Ctx250 | Combination Arm - Afa40+Ctx500
Number analyzed (Participants) | 4 | 28
ng/mL
  Cpre,ss,8 (N=4,25) | 33.2 (38.3) | 28.3 (62.3)
  Cpre,ss,15 (N=3,28) | 33.9 (19.6) | 27.1 (51.3)
  Cpre,ss,16 (N=3,0) | 36.4 (15.8) | NA (NA) — no descriptive statistics calculated due to insufficient number of participants with data
  Cpre,ss,22 (N=3,21) | 33.5 (1.30) | 28.3 (64.3)
  Cpre,ss,29 (N=3,20) | 33.4 (21.8) | 27.7 (56.8)
  Cpre,ss,43 (N=3,19) | 33.5 (14.9) | 26.0 (98.4)
  Cpre,ss,57 (N=3,0) | 36.6 (4.51) | NA (NA) — no descriptive statistics calculated due to insufficient number of participants with data

16. Secondary Outcome: Disease Control (CR, PR and Stable Disease (SD) Determined by RECIST v1.1)
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Progressive Disease (PD), At least a 20% increase in the sum of the longest diameter of target lesions or the appearance of new lesion(s); Stable Disease (SD), Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD. Disease control = CR + PR + SD.
Time Frame: up to 116 weeks
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Combination Arm - Afa40+Ctx250 | Combination Arm - Afa40+Ctx500 | Sequential Arm - Afatanib Monotherapy (Afa40 Mono) | Sequential Arm - Combination Therapy (Afa40+Ctx500)
Number analyzed (Participants) | 4 | 126 | 37 | 36
percentage of patients | 75.0 [19.4 to 99.4] | 70.6 [61.9 to 78.4] | 56.8 [39.5 to 72.9] | 50.0 [32.9 to 67.1]

17. Secondary Outcome: Objective Tumor Response (Complete Response [CR] and Partial Response [PR]) Determined by RECIST v1.1)
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Progressive Disease (PD), At least a 20% increase in the sum of the longest diameter of target lesions or the appearance of new lesion(s); Stable Disease (SD), Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD.
  Objective tumor response = CR + PR.
Time Frame: up to 116 weeks
Population: as for outcome 2
Measure: Number; unit: percentage of patients
Arm/Group | Combination Arm - Afa40+Ctx250 | Combination Arm - Afa40+Ctx500 | Sequential Arm - Afatanib Monotherapy (Afa40 Mono) | Sequential Arm - Combination Therapy (Afa40+Ctx500)
Number analyzed (Participants) | 4 | 126 | 37 | 36
percentage of patients | 0.0 | 28.6 | 5.4 | 11.1

18. Secondary Outcome: Duration of Objective Response (According to RECIST v1.1)
Description: Duration of objective response was measured from the time measurements criteria were met for CR/PR (whichever was first recorded) until the first date that recurrent or PD was objectively documented (taking as reference for PD the smallest measurements recorded since treatment started).
Time Frame: up to 116 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: months
Arm/Group | Combination Arm - Afa40+Ctx250 | Combination Arm - Afa40+Ctx500 | Sequential Arm - Afatanib Monotherapy (Afa40 Mono) | Sequential Arm - Combination Therapy (Afa40+Ctx500)
Number analyzed (Participants) | 4 | 126 | 37 | 36
months | 0 (0) | 9.00 (6.94) | 3.90 (0.07) | 5.80 (2.36)

19. Secondary Outcome: Duration of Disease Control (According to RECIST v1.1)
Description: Duration of disease control was defined as the time from the start of treatment to the time of progression or death (whichever occurred first), among patients with evidence SD, PR or CR.
Time Frame: up to 116 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: months
Arm/Group | Combination Arm - Afa40+Ctx250 | Combination Arm - Afa40+Ctx500 | Sequential Arm - Afatanib Monotherapy (Afa40 Mono) | Sequential Arm - Combination Therapy (Afa40+Ctx500)
Number analyzed (Participants) | 4 | 126 | 37 | 36
months | 7.40 (5.54) | 7.40 (5.45) | 4.90 (3.08) | 5.90 (4.51)

20. Secondary Outcome: Progression-Free Survival (PFS) Time
Description: Progression-Free Survival was defined as the duration of time from start of treatment until the day of objective tumour progression confirmed by tumour imaging (PD according to RECIST 1.1) or death.
Time Frame: up to 116 weeks
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Combination Arm - Afa40+Ctx250 | Combination Arm - Afa40+Ctx500 | Sequential Arm - Afatanib Monotherapy (Afa40 Mono) | Sequential Arm - Combination Therapy (Afa40+Ctx500)
Number analyzed (Participants) | 4 | 126 | 37 | 36
months | 4.2 [1.4 to 13.8] | 4.6 [4.2 to 6.3] | 2.7 [1.1 to 3.7] | 2.9 [1.8 to 4.8]

ADVERSE EVENTS:
Time Frame: Up to 915 days
Description: 32 patients in the 'Afa40-mono' group had disease progression and were transitioned to treatment with 'Afa40+Ctx500'. Thus the total of 203 patients (4+126+37+36) minus the 321 patients counted in both 'Afa-mono' and 'Afa40+Ctx500' treatments arms equals 171, the total number of patients started in participant flow section.
Arm/Group | Combination Arm - Afa40+Ctx250 | Combination Arm - Afa40+Ctx500 | Sequential Arm - Afatanib Monotherapy (Afa40 Mono) | Sequential Arm - Combination Therapy (Afa40+Ctx500)
Serious Adverse Events (participants affected / at risk) | 3/4 | 63/126 | 12/37 | 15/36
Other Adverse Events (participants affected / at risk) | 4/4 | 126/126 | 36/37 | 36/36
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Combination Arm - Afa40+Ctx250 (N=4) | Combination Arm - Afa40+Ctx500 (N=126) | Sequential Arm - Afatanib Monotherapy (Afa40 Mono) (N=37) | Sequential Arm - Combination Therapy (Afa40+Ctx500) (N=36)
Leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 2 | 0 | 0
Steroid withdrawal syndrome (Endocrine disorders) | 0 | 1 | 0 | 0
Diplopia (Eye disorders) | 0 | 1 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 2 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 2 | 0 | 0
Ascites (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 4 | 1 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Gastritis (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 4 | 2 | 1
Vomiting (Gastrointestinal disorders) | 0 | 6 | 3 | 1
Catheter site pain (General disorders) | 0 | 1 | 0 | 0
Chest pain (General disorders) | 1 | 1 | 1 | 0
Chills (General disorders) | 0 | 0 | 0 | 1
Death (General disorders) | 0 | 2 | 1 | 0
Fatigue (General disorders) | 0 | 3 | 0 | 0
General physical health deterioration (General disorders) | 0 | 1 | 0 | 0
Mucosal inflammation (General disorders) | 0 | 2 | 0 | 0
Oedema peripheral (General disorders) | 0 | 1 | 0 | 0
Pain (General disorders) | 0 | 2 | 0 | 0
Pyrexia (General disorders) | 0 | 2 | 0 | 2
Sudden death (General disorders) | 0 | 1 | 0 | 0
Hepatic failure (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Drug hypersensitivity (Immune system disorders) | 0 | 3 | 0 | 0
Hypersensitivity (Immune system disorders) | 0 | 1 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 1 | 0 | 0
Cystitis (Infections and infestations) | 0 | 0 | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 0 | 1 | 0
Gastroenteritis viral (Infections and infestations) | 0 | 1 | 0 | 0
Infectious pleural effusion (Infections and infestations) | 0 | 1 | 0 | 0
Meningitis aseptic (Infections and infestations) | 0 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 3 | 1 | 3
Sepsis (Infections and infestations) | 0 | 1 | 0 | 0
Streptococcal infection (Infections and infestations) | 0 | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 2 | 1 | 1
Viral infection (Infections and infestations) | 0 | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Femur fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Hip fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Spinal fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Biopsy lung (Investigations) | 0 | 1 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 5 | 2 | 0
Failure to thrive (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Spinal pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 6 | 2 | 4
Metastasis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 0 | 1
Convulsion (Nervous system disorders) | 0 | 4 | 0 | 0
Depressed level of consciousness (Nervous system disorders) | 0 | 1 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 1 | 0 | 0
Drug withdrawal headache (Nervous system disorders) | 0 | 1 | 0 | 0
Embolic cerebral infarction (Nervous system disorders) | 0 | 1 | 0 | 0
Generalised tonic-clonic seizure (Nervous system disorders) | 0 | 1 | 0 | 0
Headache (Nervous system disorders) | 0 | 1 | 0 | 0
Spinal cord compression (Nervous system disorders) | 0 | 1 | 0 | 0
Syncope (Nervous system disorders) | 0 | 2 | 0 | 1
Confusional state (Psychiatric disorders) | 0 | 1 | 0 | 0
Hallucination (Psychiatric disorders) | 0 | 0 | 0 | 1
Mental status changes (Psychiatric disorders) | 0 | 1 | 0 | 0
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 14 | 2 | 2
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 4 | 1 | 0
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 6 | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 1
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
Pain management (Surgical and medical procedures) | 0 | 1 | 0 | 0
Surgery (Surgical and medical procedures) | 0 | 1 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 2 | 0 | 1
Embolism (Vascular disorders) | 0 | 0 | 1 | 0
Hypotension (Vascular disorders) | 0 | 2 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Combination Arm - Afa40+Ctx250 (N=4) | Combination Arm - Afa40+Ctx500 (N=126) | Sequential Arm - Afatanib Monotherapy (Afa40 Mono) (N=37) | Sequential Arm - Combination Therapy (Afa40+Ctx500) (N=36)
Anaemia (Blood and lymphatic system disorders) | 0 | 5 | 2 | 3
Ear pain (Ear and labyrinth disorders) | 1 | 2 | 0 | 1
Ear pruritus (Ear and labyrinth disorders) | 1 | 1 | 0 | 0
Dry eye (Eye disorders) | 0 | 13 | 2 | 3
Eye irritation (Eye disorders) | 0 | 9 | 1 | 1
Lacrimation increased (Eye disorders) | 0 | 9 | 0 | 0
Vision blurred (Eye disorders) | 0 | 8 | 2 | 5
Abdominal pain (Gastrointestinal disorders) | 0 | 10 | 0 | 2
Abdominal pain upper (Gastrointestinal disorders) | 1 | 4 | 0 | 1
Aphthous stomatitis (Gastrointestinal disorders) | 1 | 2 | 2 | 0
Cheilitis (Gastrointestinal disorders) | 0 | 13 | 3 | 0
Constipation (Gastrointestinal disorders) | 1 | 32 | 3 | 6
Diarrhoea (Gastrointestinal disorders) | 2 | 92 | 27 | 13
Dry mouth (Gastrointestinal disorders) | 1 | 14 | 0 | 4
Glossodynia (Gastrointestinal disorders) | 1 | 5 | 1 | 2
Haemorrhoids (Gastrointestinal disorders) | 0 | 4 | 1 | 2
Large intestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Lip dry (Gastrointestinal disorders) | 0 | 1 | 2 | 1
Nausea (Gastrointestinal disorders) | 3 | 64 | 11 | 12
Oral pain (Gastrointestinal disorders) | 0 | 8 | 0 | 1
Stomatitis (Gastrointestinal disorders) | 1 | 16 | 4 | 3
Tongue ulceration (Gastrointestinal disorders) | 0 | 1 | 0 | 2
Vomiting (Gastrointestinal disorders) | 1 | 51 | 7 | 6
Asthenia (General disorders) | 0 | 7 | 1 | 3
Chest discomfort (General disorders) | 0 | 4 | 0 | 2
Chest pain (General disorders) | 2 | 6 | 1 | 2
Chills (General disorders) | 0 | 14 | 2 | 3
Face oedema (General disorders) | 1 | 0 | 0 | 0
Fatigue (General disorders) | 3 | 69 | 16 | 14
Feeling cold (General disorders) | 0 | 7 | 1 | 2
Mucosal inflammation (General disorders) | 0 | 32 | 4 | 2
Oedema peripheral (General disorders) | 0 | 12 | 3 | 4
Pain (General disorders) | 1 | 14 | 1 | 4
Pyrexia (General disorders) | 0 | 21 | 8 | 6
Xerosis (General disorders) | 0 | 53 | 0 | 0
Drug hypersensitivity (Immune system disorders) | 0 | 9 | 0 | 1
Bronchitis (Infections and infestations) | 0 | 2 | 0 | 2
Candida infection (Infections and infestations) | 0 | 3 | 0 | 2
Eye infection (Infections and infestations) | 0 | 4 | 0 | 2
Eyelid infection (Infections and infestations) | 0 | 1 | 0 | 2
Fungal infection (Infections and infestations) | 0 | 2 | 0 | 2
Impetigo (Infections and infestations) | 0 | 12 | 0 | 0
Localised infection (Infections and infestations) | 0 | 5 | 0 | 2
Nail infection (Infections and infestations) | 0 | 5 | 2 | 5
Nasopharyngitis (Infections and infestations) | 0 | 9 | 1 | 1
Paronychia (Infections and infestations) | 2 | 62 | 6 | 12
Pneumonia (Infections and infestations) | 0 | 0 | 2 | 0
Rhinitis (Infections and infestations) | 0 | 6 | 2 | 1
Skin infection (Infections and infestations) | 0 | 6 | 0 | 3
Upper respiratory tract infection (Infections and infestations) | 0 | 6 | 3 | 3
Urinary tract infection (Infections and infestations) | 0 | 11 | 5 | 6
Haemoglobin decreased (Investigations) | 0 | 3 | 0 | 2
Weight decreased (Investigations) | 1 | 10 | 5 | 4
Appetite disorder (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 2 | 28 | 7 | 8
Dehydration (Metabolism and nutrition disorders) | 0 | 2 | 2 | 5
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 1 | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 3 | 0 | 2
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 9 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 23 | 3 | 2
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 37 | 3 | 11
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 5 | 2 | 3
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 17 | 1 | 5
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 27 | 9 | 10
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 5 | 2 | 2
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 14 | 3 | 4
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 11 | 2 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 12 | 1 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 12 | 1 | 3
Pain in jaw (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0
Cognitive disorder (Nervous system disorders) | 0 | 1 | 2 | 1
Dizziness (Nervous system disorders) | 0 | 17 | 6 | 6
Dysgeusia (Nervous system disorders) | 0 | 10 | 0 | 2
Headache (Nervous system disorders) | 1 | 53 | 10 | 10
Memory impairment (Nervous system disorders) | 0 | 1 | 2 | 1
Neuropathy peripheral (Nervous system disorders) | 0 | 11 | 0 | 0
Peripheral motor neuropathy (Nervous system disorders) | 1 | 2 | 0 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 1 | 7 | 1 | 0
Anxiety (Psychiatric disorders) | 0 | 2 | 0 | 2
Depression (Psychiatric disorders) | 0 | 5 | 2 | 1
Insomnia (Psychiatric disorders) | 0 | 11 | 5 | 5
Dysuria (Renal and urinary disorders) | 1 | 9 | 0 | 0
Haemoglobinuria (Renal and urinary disorders) | 0 | 1 | 0 | 2
Pelvic pain (Reproductive system and breast disorders) | 0 | 0 | 2 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 41 | 10 | 11
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 10 | 3 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 33 | 7 | 7
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 25 | 5 | 2
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 2 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 2 | 0
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 3 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 13 | 2 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 2 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 3 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 15 | 4 | 4
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 16 | 2 | 5
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 1 | 22 | 7 | 9
Dry skin (Skin and subcutaneous tissue disorders) | 2 | 39 | 5 | 13
Erythema (Skin and subcutaneous tissue disorders) | 0 | 14 | 0 | 1
Exfoliative rash (Skin and subcutaneous tissue disorders) | 1 | 3 | 1 | 2
Hair growth abnormal (Skin and subcutaneous tissue disorders) | 0 | 3 | 0 | 3
Hirsutism (Skin and subcutaneous tissue disorders) | 0 | 17 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 1
Pain of skin (Skin and subcutaneous tissue disorders) | 0 | 10 | 0 | 0
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 0 | 8 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 50 | 1 | 6
Rash (Skin and subcutaneous tissue disorders) | 1 | 106 | 14 | 17
Rash erythematous (Skin and subcutaneous tissue disorders) | 2 | 2 | 0 | 0
Rash macular (Skin and subcutaneous tissue disorders) | 2 | 1 | 0 | 0
Skin fissures (Skin and subcutaneous tissue disorders) | 1 | 78 | 5 | 16
Skin hypertrophy (Skin and subcutaneous tissue disorders) | 0 | 2 | 2 | 0
Skin irritation (Skin and subcutaneous tissue disorders) | 0 | 7 | 0 | 1
Skin reaction (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Haematoma (Vascular disorders) | 1 | 1 | 0 | 1
Haemorrhage (Vascular disorders) | 0 | 7 | 0 | 0
Hot flush (Vascular disorders) | 1 | 0 | 0 | 0
Intra-abdominal haematoma (Vascular disorders) | 1 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any publication of the result of this trial must be consistent with the Boehringer Ingelheim publication policy. The rights of the investigator and of the sponsor with regard to publication of the results of this trial are described in the investigator contract.